CLINICAL TRIAL: NCT00890955
Title: A Phase I Study of Amrubicin and Cyclophosphamide in Patients With Advanced Solid Organ Malignancies
Brief Title: Amrubicin + Cyclophosphamide in Advanced Solid Organ Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lawrence Einhorn (Other)
Collaborators: Celgene Corporation (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Lawrence Einhorn, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG LUN07-130
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Lung Cancer
Keywords: Solid tumors
MeSH Terms: conditions — Lung Neoplasms | interventions — amrubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Amrubicin + Cyclophosphamide 3+3 design with the following dose levels:
  Dose Level -1: Amrubicin 20mg/m2, Cyclophosphamide 500mg/m2
  Dose Level 1: Amrubicin 25mg/m2, Cyclophosphamide 500mg/m2
  Dose Level 2: Amrubicin 30mg/m2, Cyclophosphamide 500mg/m2
  Dose Level 3: Amrubicin 35mg/m2, Cyclophosphamide 500mg/m2
  Dose Level 4: Amrubicin 40mg/m2, Cyclophosphamide 500mg/m2
  Interventions: Drug: Amrubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Amrubicin — * Dose Level -1: 20mg/m2
  * Dose Level 1: 25mg/m2
  * Dose Level 2: 30mg/m2
  * Dose Level 3: 35mg/m2
  * Dose Level 4: 40mg/m2
  Amrubicin will be given as a slow IV push or infusion over approximately 5 minutes once daily for 3 consecutive days starting on day 1 of each 21 day cycle.
Drug: Cyclophosphamide — Cyclophosphamide will be given at a fixed dose as 500mg/m2 IV infusion over 30-60 minutes on day 1 of each 21 day cycle (following amrubicin).

SUMMARY:
Amrubicin has shown single-agent activity in lung cancer. The combination of cyclophosphamide and anthracyclines has been studied and concluded that the combination was tolerable, could be given safely, and therapeutically useful.

This Phase I study will evaluate the combination of cyclophosphamide with amrubicin in relapsed solid tumors and will define the MTD of the combination in a US population.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

This study will follow the 3+3 design with the following dose levels:

* Dose Level -1: Amrubicin 20mg/m2, Cyclophosphamide 500mg/m2
* Dose Level 1: Amrubicin 25mg/m2, Cyclophosphamide 500mg/m2
* Dose Level 2: Amrubicin 30mg/m2, Cyclophosphamide 500mg/m2
* Dose Level 3: Amrubicin 35mg/m2, Cyclophosphamide 500mg/m2
* Dose Level 4: Amrubicin 40mg/m2, Cyclophosphamide 500mg/m2

Dose escalation starts from dose level 1.

Amrubicin will be given as a slow IV push or infusion over approximately 5 minutes once daily for 3 consecutive days starting on day 1 of each 21 day cycle.

Cyclophosphamide will be given at a fixed dose as an IV infusion over 30-60 minutes on day 1 of each 21 day cycle (following amrubicin).

ECOG Performance Status: 0-1

Life expectancy: not specified

Hematopoietic:

* Hemoglobin (Hgb) > 9 g/dL.
* Platelets > 100 K/mm3
* Absolute Neutrophil Count (ANC) > 1.5 K/mm3

Hepatic:

* Aspartate transaminase (AST) ≤ 2.5 x ULN
* Alanine transaminase (ALT) ≤ 2.5 x ULN
* Total bilirubin < 1.5 x ULN

Renal:

* Calculated creatinine clearance ≥ 60cc/min

Cardiovascular:

* Left Ventricular Ejection Fraction (LVEF) ≥ LLN for institution within 60 days prior to registration for protocol therapy.
* No history of cardiomyopathy or uncontrolled heart arrhythmia.

Pulmonary:

* No suspected, diffuse idiopathic interstitial lung disease or history of pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid organ malignancy that is refractory to currently available therapies or for which no effective therapy exists.
* Must have measurable or evaluable disease per RECIST as evaluated by imaging within 30 days prior to registration for protocol therapy.
* Must have completed chemotherapy at least 28 days prior to registration for protocol therapy and recovered from the acute toxic effects.
* Prior radiation therapy is allowed to < 25% of the bone marrow. Patients must have recovered from the acute toxic effects of radiation prior to registration for protocol therapy.
* Must be willing to consent to the blood sample collection for SNP analysis.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time of consent until at least 30 days following completion of protocol therapy.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to registration for protocol therapy. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* Written informed consent and HIPAA authorization for release of personal health information.
* Age > 18 years.

Exclusion Criteria:

* No prior therapy with cyclophosphamide or anthracyclines.
* No treatment with any investigational agent within 28 days prior to registration for protocol therapy.
* No suspected, diffuse idiopathic interstitial lung disease or history of pulmonary fibrosis.
* No evidence of severe or uncontrolled other systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.
* No symptomatic brain metastases. Patients with treated brain metastasis must be off steroids and must have completed radiation at least 21 days prior to registration for protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) of the combination of amrubicin and cyclophosphamide in patients with advanced solid tumors. | 24 months

SECONDARY OUTCOMES:
To determine the toxicities of the combination of amrubicin and cyclophosphamide in patients with advanced solid tumors. | 24 months
To assess response to the combination of amrubicin and cyclophosphamide | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Einhorn, M.D., Principal Investigator — Hoosier Cancer Research Network
Locations (10):
- United States (10):
  - Highlands Oncology Group, Springdale, Arkansas
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Siteman Cancer Center, St Louis, Missouri
  - Providence Portland Medical Center, Portland, Oregon
  - Fox Chase Cancer Center Extramural Research Program, Rockledge, Pennsylvania

REFERENCES:
- [Result] Jalal SI, Hanna N, Zon R, Masters GA, Borghaei H, Koneru K, Badve S, Prasad N, Somaiah N, Wu J, Yu Z, Einhorn L. Phase I Study of Amrubicin and Cyclophosphamide in Patients With Advanced Solid Organ Malignancies: HOG LUN 07-130. Am J Clin Oncol. 2017 Aug;40(4):329-335. doi: 10.1097/COC.0000000000000160. PMID 25503432
- See also: Hoosier Oncology Group Homepage — http://www.hoosieroncologygroup.org